CLINICAL TRIAL: NCT05176990
Title: Evaluation of the Safety of Ambulatory Surgery in Senology and Gynecology Within the Paris Saint-Joseph Hospital Group
Acronym: AMBUGYN
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: AMBUGYN
Record Dates: First submitted 2021-12-31; First posted 2022-01-04 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Ambulatory Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ambulatory surgery is defined as "surgical procedures scheduled and performed under technical conditions that imperatively require the safety of an operating room, under an anesthesia of variable mode and followed by a postoperative monitoring allowing, without increased risk, the discharge of the patient on the same day of his intervention.

It therefore does not include hospital accommodation and represents an alternative to traditional hospitalization.

Ambulatory surgery is of interest in a growing number of situations. Its interest lies on the one hand in the obvious economic interest and in the fact that this model corresponds to the expectations of patients in 2021, allowing them to return to their usual living environment as soon as possible. It also reduces the risk of infections associated with care, due to the short duration of the stay and the minimally invasive surgical techniques, without compromising safety conditions.

It therefore requires a well-designed circuit, ensuring the quality and safety of care at all stages, to allow an early return home without risk.

Since 2011, the French National Authority for Health has defined outpatient surgery as a priority objective in France, setting a target of 70% of surgeries performed as outpatient procedures by 2022.

Currently, less than 50% of surgery in France is performed on an outpatient basis, compared to 65% in Belgium, in Northern European countries and even 85% in the United States.

As early as 2001, the Assurance Maladie identified gynecological surgery as a surgery with a high potential for development in ambulatory care, particularly breast surgery and gynecological laparoscopy.

Many gynecological surgeries benefit from this type of management, in particular because of the low level of patient comorbidity, but the risks of failure are difficult to predict because of the small amount of data available in the literature, particularly in gynecology.

Paris Saint-Joseph Hospital inaugurated the Ambulatory Surgery Unit (ASU) in 2018, with a well-defined patient pathway, and outpatient surgical activity in gynecology represents 15% of activity among the 9 surgical disciplines.

The aim of this study is therefore to evaluate the safety of ambulatory management of patients operated on at the GHPSJ in the ambulatory surgery unit, in the context of breast surgery or gynaecological surgery, by assessing complications and their risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient eligible for outpatient surgery
* Patient operated in gynecology at HPSJ in UCA from 01/05/2020 to 31/05/2021
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of her data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient eligible for outpatient surgery, operated in gynecology at HPSJ in UCA from 01/05/2020 to 31/05/2021.
Sampling Method: Non-Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Complication rate of ambulatory surgery | Day 30
  This outcome corresponds to a composite criterion corresponding to the Conversion of stay to traditional hospitalization Or revision of surgery within 30 days Or re-hospitalization within 30 days Or emergency room visit within 30 days.

SECONDARY OUTCOMES:
Conversion of stay to traditional hospitalization | Day 30
  This outcome corresponds to the number of ambulatory surgery conversion of stay to traditional hospitalization.
Revision of surgery | Day 30
  This outcome corresponds to the rate of revision of surgery within 30 days.
Re-hospitalization | Day 30
  This outcome corresponds to the rate of re-hospitalization within 30 days.
Emergency room visit | Day 30
  This outcome corresponds to the rate of emergency room visit within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Severine ALRAN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Bredart A, Bottomley A, Blazeby JM, Conroy T, Coens C, D'Haese S, Chie WC, Hammerlid E, Arraras JI, Efficace F, Rodary C, Schraub S, Costantini M, Costantini A, Joly F, Sezer O, Razavi D, Mehlitz M, Bielska-Lasota M, Aaronson NK; European Organisation for Research and Treatment of Cancer Quality of Life Group and Quality of Life Unit. An international prospective study of the EORTC cancer in-patient satisfaction with care measure (EORTC IN-PATSAT32). Eur J Cancer. 2005 Sep;41(14):2120-31. doi: 10.1016/j.ejca.2005.04.041. PMID 16182120
- [Background] Marchal F, Dravet F, Classe JM, Campion L, Francois T, Labbe D, Robard S, Theard JL, Pioud R. Post-operative care and patient satisfaction after ambulatory surgery for breast cancer patients. Eur J Surg Oncol. 2005 Jun;31(5):495-9. doi: 10.1016/j.ejso.2005.01.014. PMID 15922885
- [Background] Hejl L, Raft J, Leufflen L, Rauch P, Buhler J, Abel-Decollogne F, Routiot T, Hotton J, Salleron J, Marchal F. Quality of life, anxiety, and postoperative complications of patients undergoing breast cancer surgery as ambulatory surgery compared to non-ambulatory surgery: A prospective non-randomized study. J Gynecol Obstet Hum Reprod. 2021 Feb;50(2):101779. doi: 10.1016/j.jogoh.2020.101779. Epub 2020 May 11. PMID 32407900
- [Background] Engbaek J, Bartholdy J, Hjortso NC. Return hospital visits and morbidity within 60 days after day surgery: a retrospective study of 18,736 day surgical procedures. Acta Anaesthesiol Scand. 2006 Sep;50(8):911-9. doi: 10.1111/j.1399-6576.2006.01090.x. PMID 16923084
- See also: La chirurgie du cancer du sein en ambulatoire est faisable et fiable de nos jours : étude portant sur 396 patientes — https://www.em-consulte.com/article/1097052/la-chirurgie-du-cancer-du-sein-en-ambulatoire-est-
- See also: Prise en charge ambulatoire de l'hystérectomie par voie mini-invasive : analyse des causes de résistances liées aux professionnels de santé — https://www.em-consulte.com/it/article/1333906/article/prise-en-charge-ambulatoire-de-l-hysterectomie-par